CLINICAL TRIAL: NCT02521766
Title: A Prospective, Multi-Center, Feasibility Trial of the ClarVista HARMONI™ Modular Intraocular Lens System for the Treatment of Aphakia Following Cataract Surgery
Brief Title: A Clinical Investigation of the ClarVista HARMONI™ Modular Intraocular Lens Implant Following Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ClarVista Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CP-00001
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Cataract
Keywords: Cataract; IOL; Modular IOL; IOL exchange
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- All HMIOL Cohort (Experimental): HMIOL implantation with or without optic exchange
  Interventions: Device: Harmoni Modular Intraocular Lens
- Cohort 1 (Experimental): HMIOL implantation with no optic exchange
  Interventions: Device: Harmoni Modular Intraocular Lens
- Cohort 2 (Experimental): HMIOL implantation with optic exchange
  Interventions: Device: Harmoni Modular Intraocular Lens; Procedure: Optic exchange
- Fellow Eye (Other): IOL implantation per standard of care
  Interventions: Device: Commercially Available Intraocular Lens

INTERVENTIONS:
Device: Harmoni Modular Intraocular Lens — Two-component system consisting of a base and a separate optic that allows for an intraoperative exchange of the optic only without direct manipulation of the capsular bag
  Other Names: HMIOL
  Arms: All HMIOL Cohort; Cohort 1; Cohort 2
Device: Commercially Available Intraocular Lens — IOL per investigator's standard of care
  Arms: Fellow Eye
Procedure: Optic exchange — Removal of one optic and replacement with another for the purpose of improving refractive outcomes
  Arms: Cohort 2

SUMMARY:
The main objectives of this feasibility study were:

* To demonstrate the feasibility of HARMONI Modular Intraocular Lens (HMIOL) implantation and assembly in subjects undergoing cataract surgery (All HMIOL Cohort), and
* To demonstrate the feasibility of the HMIOL optic component exchange procedure (performed 3 months following primary cataract extraction) (Cohort 2).

DETAILED DESCRIPTION:
Eligible subjects with bilateral cataracts underwent cataract extraction and IOL implantation using phacoemulsification. The study eye was implanted with the investigational device (All HMIOL Cohort). The fellow eye was treated with a commercially available intraocular lens (IOL) per standard of care procedure. At the scheduled Month 3 post-operative visit, subjects who did not opt to pursue an optic exchange procedure in the study eye were enrolled into subgroup Cohort 1 and followed for an additional 6 months. The total duration of participation for Cohort 1 was up to 15 months, which included a Day -90 to Day -1 preoperative period and a 12 month post-operative follow-up period. At the scheduled Month 3 post-operative visit, subjects who elected to pursue an optic exchange procedure in the study eye were enrolled into subgroup Cohort 2 and followed for an additional 12 months. The total duration of participation for Cohort 2 was up to 18 months, which included a Day -90 to Day -1 preoperative period, an optic exchange at Month 3 postoperative, and a 12 month post-exchange follow-up period.

Alcon Research, LLC, acquired ClarVista Medical in 2017. This study was designed and conducted by ClarVista Medical, Inc., to evaluate the safety and effectiveness of the HMIOL. The study results were collected, analyzed, and provided by ClarVista Medical, Inc. to Alcon Research, LLC.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand and provide informed consent
* Must be willing and able to return for scheduled treatment and follow-up examinations for up to 15 month study duration
* Planned bilateral removal of visually significant bilateral cataracts
* Best-corrected distance visual acuity (BCDVA) projected to be better than 20/32 after IOL implantation in both eyes
* Preoperative bilateral BCDVA of 20/40 or worse
* Both eyes must have corneal astigmatism ≤ 1.50 diopter (D)
* Women must be post-menopausal ≥1 year or surgically sterilized, or a pregnancy screen must be performed prior to the study and a reliable form of contraception, approved by the investigator, must be maintained during the study
* Dilated pupil size equal to or greater than 6 millimeters (mm) in primary study eye
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Participation in any other drug or device clinical trial within 30 days prior to enrolling in this study and/or during study participation
* History of any intraocular or corneal surgery in either eye (including refractive)
* History of any clinically significant retinal pathology or ocular diagnosis in either eye
* History of any ocular conditions which could affect the stability of the IOL
* Uncontrolled glaucoma in either eye
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. CDMA Project Lead, Surgical, Study Director — Alcon Research, LLC
Locations (2):
- ClarVista Investigational Site, Auckland, New Zealand
- ClarVista Investigational Site, Makati City, Manila, Philippines

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3 investigational sites located in the Philippines (2) and New Zealand (1).
Pre-assignment Details: Of the 217 enrolled, 101 subjects did exit the study prior to implantation, and 2 subjects failed implantation of Harmoni Modular Intraocular Lens (HMIOL). This reporting group includes all subjects with successful HMIOL implantation (114) by subgroup (Cohort 1 and Cohort 2).
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 49 | 65
Per Protocol (Successful HMIOL implantation without a major protocol deviation) | 47 | 65
Completed | 44 | 62
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Population: Per Protocol: All subjects with successful HMIOL implantation without a major protocol deviation, by subgroup (Cohort 1 and Cohort 2)
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 47 | 65 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (6.9) | 65.4 (6.7) | 66.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 40 | 71
  Male | 16 | 25 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 28 | 52 | 80
  Black | 0 | 0 | 0
  Caucasian | 19 | 11 | 30
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Postoperative BCDVA 20/40 Snellen or Better by Study Visit - All HMIOL Cohort
Description: Visual acuity (VA) was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS)-Fast method under well-lit conditions at a distance of 4 meters (m) with the correction obtained from manifest refraction testing. BCDVA was recorded in Snellen, with 20/20 considered to be 'normal' vision. A visual acuity of 20/40 means the participant is able to read a certain size letter 20 feet away that a person with 'normal' vision would be able to read from 40 feet away. This analysis was prespecified for the study eye. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 postoperative, Month 3 postoperative
Population: Per Protocol Population, with available data at the visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | All HMIOL Cohort
Number analyzed (Participants) | 112
Number analyzed (eyes) | 112
percentage of eyes
  Month 1 postoperative | 99.1
  Month 3 postoperative | 100.0

2. Primary Outcome: Percentage of Eyes With Postoperative BCDVA 20/40 Snellen or Better by Study Visit - Cohort 1
Description: VA was assessed using the ETDRS-Fast method under well-lit conditions at a distance of 4 m with the correction obtained from manifest refraction testing. BCDVA was recorded in Snellen, with 20/20 considered to be 'normal' vision. A visual acuity of 20/40 means the participant is able to read a certain size letter 20 feet away that a person with 'normal' vision would be able to read from 40 feet away. This analysis was prespecified for the study eye. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 postoperative, Month 3 postoperative, Month 6 postoperative, Month 12 postoperative
Population: Per Protocol Population, with available data at the visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Cohort 1
Number analyzed (Participants) | 47
Number analyzed (eyes) | 47
percentage of eyes
  Month 1 postoperative | 100.0
  Month 3 postoperative | 100.0
  Month 6 postoperative | 100.0
  Month 12 postoperative: number analyzed (Participants) | 43
  Month 12 postoperative: number analyzed (eyes) | 43
  Month 12 postoperative | 100.0

3. Primary Outcome: Percentage of Eyes With Postoperative BCDVA 20/40 Snellen or Better by Study Visit - Cohort 2
Description: VA was assessed using the ETDRS-Fast method under well-lit conditions at a distance of 4 m with the correction obtained from manifest refraction testing. BCDVA was recorded in Snellen, with 20/20 considered to be 'normal' vision. A visual acuity of 20/40 means the participant is able to read a certain size letter 20 feet away that a person with 'normal' vision would be able to read from 40 feet away. An optic exchange occurred at the Month 3 visit, after which subjects were followed for an additional 12 months. Month 1 postoperative and Month 3 postoperative visits were pre-optic exchange. This analysis was prespecified for the study eye. No formal statistical hypothesis testing was planned
Time Frame: Month 1 postoperative, Month 3 postoperative, Week 1 post-optic exchange, Month 1 post-optic exchange, Month 3 post-optic exchange, Month 6 post-optic exchange, Month 12 post-optic exchange
Population: Per Protocol Population, with available data at the visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Cohort 2
Number analyzed (Participants) | 65
Number analyzed (eyes) | 65
percentage of eyes
  Month 1 postoperative | 98.5
  Month 3 postoperative | 100
  Week 1 post-optic exchange | 100
  Month 1 post-optic exchange: number analyzed (Participants) | 64
  Month 1 post-optic exchange: number analyzed (eyes) | 64
  Month 1 post-optic exchange | 100
  Month 3 post-optic exchange: number analyzed (Participants) | 63
  Month 3 post-optic exchange: number analyzed (eyes) | 63
  Month 3 post-optic exchange | 100
  Month 6 post-optic exchange: number analyzed (Participants) | 63
  Month 6 post-optic exchange: number analyzed (eyes) | 63
  Month 6 post-optic exchange | 100
  Month 12 post-optic exchange: number analyzed (Participants) | 62
  Month 12 post-optic exchange: number analyzed (eyes) | 62
  Month 12 post-optic exchange | 96.8

4. Primary Outcome: Percentage of Eyes With Postoperative BCDVA 20/40 Snellen or Better by Study Visit - Fellow Eye
Description: as for outcome 2
Time Frame: Month 1 postoperative, Month 3 postoperative, Month 12 postoperative
Population: Per Protocol Population, with available data at the visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Fellow Eye
Number analyzed (Participants) | 111
Number analyzed (eyes) | 111
percentage of eyes
  Month 1 postoperative: number analyzed (Participants) | 106
  Month 1 postoperative: number analyzed (eyes) | 106
  Month 1 postoperative | 100.0
  Month 3 postoperative | 100.0
  Month 12 postoperative: number analyzed (Participants) | 108
  Month 12 postoperative: number analyzed (eyes) | 108
  Month 12 postoperative | 100.0

5. Primary Outcome: Percentage of Eyes With Postoperative Manifest Refraction Spherical Equivalent (MRSE) Within Target by Study Visit - All HMIOL Cohort
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. The manifest refraction spherical equivalent (MRSE) was calculated as follows: sphere + 1/2 cylinder, and measured in diopters (D). This analysis was prespecified for the study eye. No formal statistical hypothesis testing was planned.
Time Frame: Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: Per Protocol Population, with available data at the visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | All HMIOL Cohort
Number analyzed (Participants) | 112
Number analyzed (eyes) | 112
percentage of eyes
  Week 1 postoperative: Within ± 0.5 D of Target: number analyzed (Participants) | 109
  Week 1 postoperative: Within ± 0.5 D of Target: number analyzed (eyes) | 109
  Week 1 postoperative: Within ± 0.5 D of Target | 33.9
  Week 1 postoperative: Within ± 1.0 D of Target: number analyzed (Participants) | 109
  Week 1 postoperative: Within ± 1.0 D of Target: number analyzed (eyes) | 109
  Week 1 postoperative: Within ± 1.0 D of Target | 70.6
  Month 1 postoperative: Within ± 0.5 D of Target | 26.8
  Month 1 postoperative: Within ± 1.0 D of Target | 61.6
  Month 3 postoperative: Within ± 0.5 D of Target | 19.6
  Month 3 postoperative: Within ± 1.0 D of Target | 52.7

6. Primary Outcome: Percentage of Eyes With Postoperative Manifest Refraction Spherical Equivalent (MRSE) Within Target by Study Visit - Cohort 1
Description: as for outcome 5
Time Frame: Week 1 postoperative, Month 1 postoperative, Month 3 postoperative, Month 6 postoperative, Month 12 postoperative
Population: Per Protocol Population, with available data at the visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Cohort 1
Number analyzed (Participants) | 47
Number analyzed (eyes) | 47
percentage of eyes
  Week 1 postoperative: Within ± 0.5 D of Target: number analyzed (Participants) | 45
  Week 1 postoperative: Within ± 0.5 D of Target: number analyzed (eyes) | 45
  Week 1 postoperative: Within ± 0.5 D of Target | 31.1
  Week 1 postoperative: Within ± 1.0 D of Target: number analyzed (Participants) | 45
  Week 1 postoperative: Within ± 1.0 D of Target: number analyzed (eyes) | 45
  Week 1 postoperative: Within ± 1.0 D of Target | 57.8
  Month 1 postoperative: Within ± 0.5 D of Target | 23.4
  Month 1 postoperative: Within ± 1.0 D of Target | 48.9
  Month 3 postoperative: Within ± 0.5 D of Target | 19.1
  Month 3 postoperative: Within ± 1.0 D of Target | 44.7
  Month 6 postoperative: Within ± 0.5 D of Target | 14.9
  Month 6 postoperative: Within ± 1.0 D of Target | 44.7
  Month 12 postoperative: Within ± 0.5 D of Target: number analyzed (Participants) | 43
  Month 12 postoperative: Within ± 0.5 D of Target: number analyzed (eyes) | 43
  Month 12 postoperative: Within ± 0.5 D of Target | 20.9
  Month 12 postoperative: Within ± 1.0 D of Target: number analyzed (Participants) | 43
  Month 12 postoperative: Within ± 1.0 D of Target: number analyzed (eyes) | 43
  Month 12 postoperative: Within ± 1.0 D of Target | 37.2

7. Primary Outcome: Percentage of Eyes With Postoperative Manifest Refraction Spherical Equivalent (MRSE) Within Target by Study Visit - Cohort 2
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. The manifest refraction spherical equivalent (MRSE) was calculated as follows: sphere + 1/2 cylinder, and measured in diopters (D). An optic exchange occurred at the Month 3 visit, after which subjects were followed for an additional 12 months. Week 1 postoperative, Month 1 postoperative, and Month 3 postoperative visits were pre-optic exchange. This analysis was prespecified for the study eye. No formal statistical hypothesis testing was planned.
Time Frame: Week 1 postoperative, Month 1 postoperative, Month 3 postoperative, Week 1 post-optic exchange, Month 1 post-optic exchange, Month 3 post-optic exchange, Month 6 post-optic exchange, Month 12 post-optic exchange
Population: Per Protocol Population, with available data at the visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Cohort 2
Number analyzed (Participants) | 65
Number analyzed (eyes) | 65
percentage of eyes
  Week 1 postoperative: Within ± 0.5 D of Target: number analyzed (Participants) | 64
  Week 1 postoperative: Within ± 0.5 D of Target: number analyzed (eyes) | 64
  Week 1 postoperative: Within ± 0.5 D of Target | 35.9
  Week 1 postoperative: Within ± 1.0 D of Target: number analyzed (Participants) | 64
  Week 1 postoperative: Within ± 1.0 D of Target: number analyzed (eyes) | 64
  Week 1 postoperative: Within ± 1.0 D of Target | 79.7
  Month 1 postoperative: Within ± 0.5 D of Target | 29.2
  Month 1 postoperative: Within ± 1.0 D of Target | 70.8
  Month 3 postoperative: Within ± 0.5 D of Target | 20.0
  Month 3 postoperative: Within ± 1.0 D of Target | 58.5
  Week 1 post-exchange: Within ± 0.5 D of Target | 76.9
  Week 1 post-exchange: Within ± 1.0 D of Target | 98.5
  Month 1 post-exchange: Within ± 0.5 D of Target: number analyzed (Participants) | 64
  Month 1 post-exchange: Within ± 0.5 D of Target: number analyzed (eyes) | 64
  Month 1 post-exchange: Within ± 0.5 D of Target | 82.8
  Month 1 post-exchange: Within ± 1.0 D of Target: number analyzed (Participants) | 64
  Month 1 post-exchange: Within ± 1.0 D of Target: number analyzed (eyes) | 64
  Month 1 post-exchange: Within ± 1.0 D of Target | 100.0
  Month 3 post-exchange: Within ± 0.5 D of Target: number analyzed (Participants) | 63
  Month 3 post-exchange: Within ± 0.5 D of Target: number analyzed (eyes) | 63
  Month 3 post-exchange: Within ± 0.5 D of Target | 81.0
  Month 3 post-exchange: Within ± 1.0 D of Target: number analyzed (Participants) | 63
  Month 3 post-exchange: Within ± 1.0 D of Target: number analyzed (eyes) | 63
  Month 3 post-exchange: Within ± 1.0 D of Target | 98.4
  Month 6 post-exchange: Within ± 0.5 D of Target: number analyzed (Participants) | 63
  Month 6 post-exchange: Within ± 0.5 D of Target: number analyzed (eyes) | 63
  Month 6 post-exchange: Within ± 0.5 D of Target | 84.1
  Month 6 post-exchange: Within ± 1.0 D of Target: number analyzed (Participants) | 63
  Month 6 post-exchange: Within ± 1.0 D of Target: number analyzed (eyes) | 63
  Month 6 post-exchange: Within ± 1.0 D of Target | 100.0
  Month 12 post-exchange: Within ± 0.5 D of Target: number analyzed (Participants) | 62
  Month 12 post-exchange: Within ± 0.5 D of Target: number analyzed (eyes) | 62
  Month 12 post-exchange: Within ± 0.5 D of Target | 77.4
  Month 12 post-exchange: Within ± 1.0 D of Target: number analyzed (Participants) | 62
  Month 12 post-exchange: Within ± 1.0 D of Target: number analyzed (eyes) | 62
  Month 12 post-exchange: Within ± 1.0 D of Target | 95.2

8. Primary Outcome: Percentage of Eyes With Postoperative Manifest Refraction Spherical Equivalent (MRSE) Within Target by Study Visit - Fellow Eye
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. The manifest refraction spherical equivalent (MRSE) was calculated as follows: sphere + 1/2 cylinder, and measured in diopters (D). This analysis was prespecified for the fellow eye. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 postoperative, Month 3 postoperative, Month 12 postoperative
Population: Per Protocol Population, with available data at the visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Fellow Eye
Number analyzed (Participants) | 111
Number analyzed (eyes) | 111
percentage of eyes
  Month 1 postoperative: Within ± 0.5 D of Target: number analyzed (Participants) | 107
  Month 1 postoperative: Within ± 0.5 D of Target: number analyzed (eyes) | 107
  Month 1 postoperative: Within ± 0.5 D of Target | 78.5
  Month 1 postoperative: Within ± 1.0 D of Target: number analyzed (Participants) | 107
  Month 1 postoperative: Within ± 1.0 D of Target: number analyzed (eyes) | 107
  Month 1 postoperative: Within ± 1.0 D of Target | 98.1
  Month 3 postoperative: Within ± 0.5 D of Target | 81.1
  Month 3 postoperative: Within ± 1.0 D of Target | 99.1
  Month 12 postoperative: Within ± 0.5 D of Target: number analyzed (Participants) | 108
  Month 12 postoperative: Within ± 0.5 D of Target: number analyzed (eyes) | 108
  Month 12 postoperative: Within ± 0.5 D of Target | 72.2
  Month 12 postoperative: Within ± 1.0 D of Target: number analyzed (Participants) | 108
  Month 12 postoperative: Within ± 1.0 D of Target: number analyzed (eyes) | 108
  Month 12 postoperative: Within ± 1.0 D of Target | 97.2

9. Primary Outcome: Mean BCDVA (Letters Read) by Study Visit - All HMIOL Cohort
Description: VA was assessed using the ETDRS-Fast method under well-lit conditions at a distance of 4 m with the correction obtained from manifest refraction testing. BCDVA was recorded in letters read correctly. This analysis was prespecified for the study eye. No formal statistical hypothesis testing was planned.
Time Frame: Day -90 to Day -1 preoperative, Month 1 postoperative, Month 3 postoperative
Population: Per Protocol Population, with available data at the visit
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | All HMIOL Cohort
Number analyzed (Participants) | 112
Number analyzed (eyes) | 112
letters
  Day -90 to Day -1 preoperative | 75.2 (14.2)
  Month 1 postoperative | 84.6 (4.5)
  Month 3 postoperative | 85.4 (3.8)

10. Primary Outcome: Mean BCDVA (Letters Read) by Study Visit - Cohort 1
Description: as for outcome 9
Time Frame: Day -90 to -1 preoperative, Month 1 postoperative, Month 3 postoperative, Month 6 postoperative, Month 12 postoperative
Population: Per Protocol Population, with available data at the visit
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | Cohort 1
Number analyzed (Participants) | 47
Number analyzed (eyes) | 47
letters
  Day -90 to -1 preoperative | 79.9 (9.4)
  Month 1 postoperative | 85.8 (3.6)
  Month 3 postoperative | 86.7 (3.5)
  Month 6 postoperative | 86.2 (3.9)
  Month 12 postoperative: number analyzed (Participants) | 43
  Month 12 postoperative: number analyzed (eyes) | 43
  Month 12 postoperative | 86.2 (4.5)

11. Primary Outcome: Mean BCDVA (Letters Read) by Study Visit - Cohort 2
Description: VA was assessed using the ETDRS-Fast method under well-lit conditions at a distance of 4 m with the correction obtained from manifest refraction testing. BCDVA was recorded in letters read correctly. An optic exchange occurred at the Month 3 visit, after which subjects were followed for an additional 12 months. Month 1 postoperative and Month 3 postoperative visits were pre-optic exchange.This analysis was prespecified for the study eye. No formal statistical hypothesis testing was planned.
Time Frame: Day -90 to -1 preoperative, Month 1 postoperative, Month 3 postoperative, Week 1 post-optic exchange, Month 1 post-optic exchange, Month 3 post-optic exchange, Month 6 post-optic exchange, Month 12 post-optic exchange
Population: Per Protocol Population, with available data at the visit
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | Cohort 2
Number analyzed (Participants) | 65
Number analyzed (eyes) | 65
letters
  Day -90 to -1 preoperative | 71.8 (16.1)
  Month 1 postoperative | 83.7 (4.9)
  Month 3 postoperative | 84.4 (3.8)
  Week 1 post-optic exchange | 84.5 (4.4)
  Month 1 post-optic exchange: number analyzed (Participants) | 64
  Month 1 post-optic exchange: number analyzed (eyes) | 64
  Month 1 post-optic exchange | 85.1 (4.0)
  Month 3 post-optic exchange: number analyzed (Participants) | 63
  Month 3 post-optic exchange: number analyzed (eyes) | 63
  Month 3 post-optic exchange | 85.2 (4.0)
  Month 6 post-optic exchange: number analyzed (Participants) | 63
  Month 6 post-optic exchange: number analyzed (eyes) | 63
  Month 6 post-optic exchange | 85.6 (3.5)
  Month 12 post-optic exchange: number analyzed (Participants) | 62
  Month 12 post-optic exchange: number analyzed (eyes) | 62
  Month 12 post-optic exchange | 83.5 (9.9)

12. Primary Outcome: Mean BCDVA (Letters Read) by Study Visit - Fellow Eye
Description: VA was assessed using the ETDRS-Fast method under well-lit conditions at a distance of 4 m with the correction obtained from manifest refraction testing. BCDVA was rrecorded in letters read correctly. This analysis was prespecified for the fellow eye. No formal statistical hypothesis testing was planned.
Time Frame: Day -90 to -1 preoperative, Month 1 postoperative, Month 3 postoperative, Month 12 postoperative
Population: Per Protocol Population, with available data at the visit
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | Fellow Eye
Number analyzed (Participants) | 114
Number analyzed (eyes) | 114
letters
  Day -90 to -1 preoperative | 74.5 (17.9)
  Month 1 postoperative: number analyzed (Participants) | 106
  Month 1 postoperative: number analyzed (eyes) | 106
  Month 1 postoperative | 86.3 (4.0)
  Month 3 postoperative: number analyzed (Participants) | 111
  Month 3 postoperative: number analyzed (eyes) | 111
  Month 3 postoperative | 86.9 (3.4)
  Month 12 postoperative: number analyzed (Participants) | 108
  Month 12 postoperative: number analyzed (eyes) | 108
  Month 12 postoperative | 86.9 (3.5)

13. Primary Outcome: Mean Uncorrected Distance Visual Acuity (UCDVA) (Letters Read) by Study Visit - All HMIOL Cohort
Description: VA was assessed using the ETDRS-Fast method under well-lit conditions at a distance of 4 m with an optical infinity adjustment of +0.25 diopter (D). UCDVA was recorded in letters read correctly. This analysis was prespecified for the study eye. No formal statistical hypothesis testing was planned.
Time Frame: Day 1 postoperative, Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: Per Protocol Population, with available data at the visit
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | All HMIOL Cohort
Number analyzed (Participants) | 112
Number analyzed (eyes) | 112
letters
  Day 1 postoperative: number analyzed (Participants) | 111
  Day 1 postoperative: number analyzed (eyes) | 111
  Day 1 postoperative | 71.5 (11.0)
  Week 1 postoperative: number analyzed (Participants) | 111
  Week 1 postoperative: number analyzed (eyes) | 111
  Week 1 postoperative | 70.4 (10.1)
  Month 1 postoperative | 70.6 (10.2)
  Month 3 postoperative | 73.4 (9.3)

14. Primary Outcome: Mean Uncorrected Distance Visual Acuity (UCDVA) (Letters Read) by Study Visit - Cohort 1
Description: as for outcome 13
Time Frame: Day 1 postoperative, Week 1 postoperative, Month 1 postoperative, Month 3 postoperative, Month 6 postoperative, Month 12 postoperative
Population: Per Protocol Population, with available data at the visit
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | Cohort 1
Number analyzed (Participants) | 47
Number analyzed (eyes) | 47
letters
  Day 1 postoperative | 74.8 (10.2)
  Week 1 postoperative | 73.7 (9.2)
  Month 1 postoperative | 75.4 (8.3)
  Month 3 postoperative | 77.1 (8.2)
  Month 6 postoperative | 78.1 (7.3)
  Month 12 postoperative: number analyzed (Participants) | 43
  Month 12 postoperative: number analyzed (eyes) | 43
  Month 12 postoperative | 77.9 (6.9)

15. Primary Outcome: Mean Uncorrected Distance Visual Acuity (UCDVA) (Letters Read) by Study Visit - Cohort 2
Description: VA was assessed using the ETDRS-Fast method under well-lit conditions at a distance of 4 m with an optical infinity adjustment of +0.25 diopter (D). UCDVA was recorded in letters read correctly. An optic exchange occurred at the Month 3 visit, after which subjects were followed for an additional 12 months. Day 1 postoperative, Week 1 postoperative, Month 1 postoperative, and Month 3 postoperative visits were pre-optic exchange. This analysis was prespecified for the study eye. No formal statistical hypothesis testing was planned.
Time Frame: Day 1 postoperative, Week 1 postoperative, Month 1 postoperative, Month 3 postoperative, Day 1 post-optic exchange, Week 1 post-optic exchange, Month 1 post-optic exchange, Month 3 post-optic exchange, Month 6 post-optic exchange, Month 12 post-optic exch
Population: Per Protocol Population, with available data at the visit
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | Cohort 2
Number analyzed (Participants) | 65
Number analyzed (eyes) | 65
letters
  Day 1 postoperative | 69.1 (10.9)
  Week 1 postoperative | 68.1 (10.2)
  Month 1 postoperative | 67.2 (10.2)
  Month 3 postoperative | 70.7 (9.2)
  Day 1 post-optic exchange | 76.8 (13.4)
  Week 1 post-optic exchange | 79.8 (6.0)
  Month 1 post-optic exchange: number analyzed (Participants) | 64
  Month 1 post-optic exchange: number analyzed (eyes) | 64
  Month 1 post-optic exchange | 80.7 (6.4)
  Month 3 post-optic exchange: number analyzed (Participants) | 63
  Month 3 post-optic exchange: number analyzed (eyes) | 63
  Month 3 post-optic exchange | 81.1 (5.5)
  Month 6 post-optic exchange: number analyzed (Participants) | 63
  Month 6 post-optic exchange: number analyzed (eyes) | 63
  Month 6 post-optic exchange | 81.2 (5.4)
  Month 12 post-optic exchange: number analyzed (Participants) | 62
  Month 12 post-optic exchange: number analyzed (eyes) | 62
  Month 12 post-optic exchange | 78.2 (13.4)

16. Primary Outcome: Mean Uncorrected Distance Visual Acuity (UCDVA) (Letters Read) by Study Visit - Fellow Eye
Description: VA was assessed using the ETDRS-Fast method under well-lit conditions at a distance of 4 m with an optical infinity adjustment of +0.25 diopter (D). UCDVA was recorded in letters read correctly. This analysis was prespecified for the fellow eye. No formal statistical hypothesis testing was planned.
Time Frame: as for outcome 14
Population: Per Protocol Population, with available data at the visit
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | Fellow Eye
Number analyzed (Participants) | 114
Number analyzed (eyes) | 114
letters
  Day 1 postoperative: number analyzed (Participants) | 111
  Day 1 postoperative: number analyzed (eyes) | 111
  Day 1 postoperative | 80.6 (8.0)
  Week 1 postoperative | 81.3 (6.4)
  Month 1 postoperative | 81.3 (5.8)
  Month 3 postoperative: number analyzed (Participants) | 111
  Month 3 postoperative: number analyzed (eyes) | 111
  Month 3 postoperative | 82.4 (5.4)
  Month 6 postoperative: number analyzed (Participants) | 107
  Month 6 postoperative: number analyzed (eyes) | 107
  Month 6 postoperative | 83.0 (5.0)
  Month 12 postoperative: number analyzed (Participants) | 108
  Month 12 postoperative: number analyzed (eyes) | 108
  Month 12 postoperative | 82.1 (5.5)

17. Primary Outcome: Percentage of Eyes With UCDVA by Category (Snellen) for Each Post-optic Exchange Study Visit - Cohort 2
Description: VA was assessed using the ETDRS-Fast method under well-lit conditions at a distance of 4 m with an optical infinity adjustment of +0.25 diopter (D). UCDVA was recorded in Snellen, with 20/20 considered to be 'normal' vision. A visual acuity of 20/40 means the participant is able to read a certain size letter 20 feet away that a person with 'normal' vision would be able to read from 40 feet away. An optic exchange occurred at the Month 3 visit, after which subjects were followed for an additional 12 months. Day 1 postoperative, Week 1 postoperative, Month 1 postoperative, and Month 3 postoperative visits were pre-optic exchange. This analysis was prespecified for the study eye, Cohort 2 only. No formal statistical hypothesis testing was planned.
Time Frame: Day 1 post-optic exchange, Week 1 post-optic exchange, Month 1 post-optic exchange, Month 3 post-optic exchange, Month 6 post-optic exchange, Month 12 post-optic exchange
Population: Per Protocol Population, with available data at the visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Cohort 2 Day 1 Post-optic Exchange; Cohort 2 Week 1 Post-optic Exchange; Cohort 2 Month 1 Post-optic Exchange; Cohort 2 Month 3 Post-optic Exchange; Cohort 2 Month 6 Post-optic Exchange; Cohort 2 Month 12 Post-optic Exchange: HMIOL implantation with optic exchange
Arm/Group | Cohort 2 Day 1 Post-optic Exchange | Cohort 2 Week 1 Post-optic Exchange | Cohort 2 Month 1 Post-optic Exchange | Cohort 2 Month 3 Post-optic Exchange | Cohort 2 Month 6 Post-optic Exchange | Cohort 2 Month 12 Post-optic Exchange
Number analyzed (Participants) | 65 | 65 | 64 | 63 | 63 | 62
Number analyzed (eyes) | 65 | 65 | 64 | 63 | 63 | 63
percentage of eyes
  20/20 Snellen or Better | 41.5 | 47.7 | 53.1 | 49.2 | 55.6 | 50.0
  20/25 Snellen or Better | 67.7 | 69.2 | 70.3 | 81.0 | 79.4 | 74.2
  20/32 Snellen or Better | 80.0 | 87.7 | 92.2 | 93.7 | 93.7 | 83.9
  20/40 Snellen or Better | 87.7 | 93.8 | 96.9 | 96.8 | 98.4 | 95.2
  Worse than 20/40 Snellen | 12.3 | 6.2 | 3.1 | 3.2 | 1.6 | 4.8

18. Primary Outcome: Mesopic Best Corrected Distance Visual Acuity (mBCDVA) (With and Without Glare) (Letters Read) at Study Visit - All HMIOL Cohort
Description: VA was assessed using the ETDRS-Fast method under mesopic (dimly lit) conditions at a distance of 4 m with the correction obtained from manifest refraction testing. Testing was performed with and without glare. Chart luminance was set to 3 cd/m2. mBCDVA was recorded in letters read correctly. This analysis was prespecified for the study eye, All HMIOL Cohort only. No formal statistical hypothesis testing was planned.
Time Frame: Month 3 postoperative
Population: Per Protocol Population, with available data at the visit
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: eyes
Arm/Group | All HMIOL Cohort
Number analyzed (Participants) | 112
Number analyzed (eyes) | 112
letters
  With glare | 81.0 (4.9)
  Without glare | 81.1 (5.6)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent until study: Cohort 1: Up to 15 months, including a Day -90 to Day -1 preoperative period and a 12 month post-operative follow-up period. Cohort 2: Up to 18 months, including a Day -90 to Day -1 preoperative period, an optic exchange at Month 3 postoperative, and a 12 month post-exchange follow-up period. "At Risk" population of systemic AEs is reported in units of subjects; all other AE populations are reported in units of eyes.
Description: Safety Analysis Population: All eyes with attempted study lens (HMIOL) implantation (successful or aborted after contact with the eye).
Groups:
- Cohort 1 (Ocular): HMIOL implantation with no optic exchange
  Events reported in this group occurred in the study eye from time of consent to study exit (up to 15 months)
- Cohort 2 Pre-exchange (Ocular): HMIOL implantation pre-optic exchange
  Events reported in this group occurred in the study eye from time of consent to time of optic exchange (up to 6 months)
- Cohort 2 Post-exchange (Ocular): HMIOL implantation post-optic exchange
  Events reported in this group occurred in the study eye from time of optic exchange to time of study exit (up to 12 months)
- Fellow Eye (Ocular): IOL per standard of care
  Events reported in this group occurred in the fellow eye from time of consent to study exit (up to 15 months if study eye was enrolled in Cohort 1, up to 18 months if study eye was enrolled in Cohort 2)
- Systemic (Non-ocular): Events reported in this group occurred from time of consent to study exit (up to 15 months if subject was enrolled in Cohort 1, up to 18 months if subject was enrolled in Cohort 2)
Arm/Group | Cohort 1 (Ocular) | Cohort 2 Pre-exchange (Ocular) | Cohort 2 Post-exchange (Ocular) | Fellow Eye (Ocular) | Systemic (Non-ocular)
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/65 | 0/65 | 0/114 | 0/114
Serious Adverse Events (participants affected / at risk) | 2/51 | 2/65 | 0/65 | 2/114 | 4/114
Other Adverse Events (participants affected / at risk) | 2/51 | 1/65 | 6/65 | 5/114 | 0/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Ocular) (N=51) | Cohort 2 Pre-exchange (Ocular) (N=65) | Cohort 2 Post-exchange (Ocular) (N=65) | Fellow Eye (Ocular) (N=114) | Systemic (Non-ocular) (N=114)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Endophthalmitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Neovascular age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 1 | 0
Posterior Capsule Rupture (Eye disorders) | 1 | 0 | 0 | 0 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Parkinsonism (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Eye operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Intraocular lens implant (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Ocular) (N=51) | Cohort 2 Pre-exchange (Ocular) (N=65) | Cohort 2 Post-exchange (Ocular) (N=65) | Fellow Eye (Ocular) (N=114) | Systemic (Non-ocular) (N=114)
Dry eye (Eye disorders) | 2 | 1 | 6 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2016-03-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT02521766/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT02521766/SAP_001.pdf